CLINICAL TRIAL: NCT00652197
Title: A Flow Monitor for Pediatric Hydrocephalic Shunts - Flow Sensor Study
Brief Title: Monitoring Patient Cerebro-Spinal Fluid Drainage With an Ultrasonic Flow Sensor
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-HYDRO-1A-H; 2R44NS049680-02 (NIH)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; shunt dysfunction; shunt flow
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extraventricular Drainage: Includes pediatric hydrocephalus patients that are in recovery from shunt explanation.

SUMMARY:
The study hypothesis is that an ultrasonic flow sensor can accurately measure flow in hydrocephalic shunts.

The ultrasonic sensor will measure cerebro-spinal fluid drainage in hydrocephalus patients with external ventriculostomies and extra-ventricular drainage systems. The sensor measurements will be compared with the volume of fluid collected by the drainage bag.

After a 24-hour measurement period, the doctor will change the drainage bag position to simulate the patient sitting up and leaning back, to see if this temporarily stops flow through the drainage line.

This data will show whether the sensor accurately measures typical drainage flows seen in hydrocephalus patients. This research will help develop an implantable flow monitor for pediatric hydrocephalus patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: newborn through age 20
* Diagnosed with Hydrocephalus
* Instrumented with an Extra-Ventricular Drainage Line

Exclusion Criteria:

* Age: older than age 20
* Not diagnosed with Hydrocephalus
* Not instrumented with an Extra-Ventricular Drainage Line

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hydrocephalus patients under the care of the Children's Hospital of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage system. | 24-hour period

SECONDARY OUTCOMES:
Recording of the pressure waveform related to the volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage system. | 24-hour period

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J Drost, BS, MS, Principal Investigator — Transonic Systems Inc.; Bruce A Kaufman, MD, Study Director — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States